CLINICAL TRIAL: NCT02174692
Title: Exploring the Metabolic and Molecular Basis of Age-related Declines in Human Skeletal Muscle Regenerative Capacity
Brief Title: Study of Muscle Repair Following Exercise in Young and Elderly People
Acronym: MDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MDS
Record Dates: First submitted 2014-06-11; First posted 2014-06-25 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Elderly (Experimental): Exercise One leg eccentric exercise: 7 sets of 10 repetitions at 80% 1 repetition maximum Contralateral leg concentric exercise: 7 sets of 10 repetitions at 80% 1 repetition maximum
  2 minutes rest between sets
  Interventions: Other: Exercise
- Young (Experimental): Exercise
  One leg eccentric exercise: 7 sets of 10 repetitions at 80% 1 repetition maximum Contralateral leg concentric exercise: 7 sets of 10 repetitions at 80% 1 repetition maximum
  2 minutes rest between sets
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — One leg eccentric exercise: 7 sets of 10 repetitions at 80% 1 repetition maximum Contralateral leg concentric exercise: 7 sets of 10 repetitions at 80% 1 repetition maximum
  2 mins rest between sets

SUMMARY:
The aim of this study is to understand how healthy muscle repairs in response to eccentric exercise by evaluating functional, metabolic and molecular measures. Furthermore, this study will aim to understand the repair mechanisms in elderly healthy muscle following eccentric exercise by evaluating the same measures and highlighting age-related differences in repair mechanisms which may account for the age-related loss in muscle mass. It is hypothesised that elderly muscle will have a lesser/ blunted repair process compared to young muscle.

To meet the aims of this study and to answer the hypothesis, this study protocol is as follows:

Baseline functional, metabolic and molecular values are obtained via functional testing and a muscle biopsy. Participants then perform eccentric exercise designed to induce functional decline and muscle soreness and the contralateral leg performs concentric exercise which isn't designed to induce soreness or functional decline. Using a time-course, various metabolic and molecular measures are taken prior to and up to 7 days post exercise to understand the mechanisms underlying muscle repair. In addition the use of a novel amino acid tracer (D2O) will allow for synthesis measures over the duration of the study rather than the typical tracer techniques which only capture ~12 hours of synthesis.

DETAILED DESCRIPTION:
Participation in this study requires participants to attend the laboratory fasted on 5 occasions spread over a period of 12 days.

Participants will report to the laboratory on the first visit for a blood sample and muscle biopsy. In order to measure muscle metabolism participants will also consume 'heavy water', which will also require participants to provide daily saliva swabs.

After 96 hours participants will be asked to arrive at the laboratory to perform a bout of heavy exercise on one leg to induce sensations of muscle soreness in the days following exercise. Investigators will then collect a blood sample and muscle biopsy from the exercised leg and do exercise tests. After this, participants will perform another bout of exercise on the other leg that will also be followed immediately by a blood sample, muscle biopsy and exercise tests. This second exercise bout is not designed to induce sensations of muscle soreness. After 5 hours , exercise tests will be performed and a further blood sample and biopsies from both legs will be collected.

Approximately, 21 hours after exercise (visit 3) participants will be asked to return to the lab for a short infusion (2.5 hour duration) of 2-deoxyglucose (2DOG), which allows investigators to measure glucose uptake. After the infusion, a blood and a muscle biopsy will be taken from each leg followed by exercising testing. Participants will then report back to the laboratory for exercise testing, a blood sample and a single muscle biopsy from both legs at 72 (visit 4) and 168 hours (visit 5) after the initial exercise session.

ELIGIBILITY:
Inclusion Criteria:

* 16-30 kg/m2 BMI
* Male
* Sedentary
* 18-28 years or 65-75 years

Exclusion Criteria:

* Active cardiovascular disease
* Cerebrovascular disease including previous stroke or aneurysm
* Respiratory disease including pulmonary hypertension or chronic obstructive pulmonary disease
* Metabolic disease including:

  * hyper/ hypo parathyroidism or thyroidism
  * Cushing's disease
  * Type 1 or 2 diabetes
* Active inflammatory bowel disease
* Renal disease
* Malignancy
* Recent steroid treatment (within 6 months), or hormone replacement therapy
* Clotting dysfunction
* Musculoskeletal or neurological disorders medication that affects muscle metabolism ie. paracetamol or non steroidal anti inflammatories (NSAID's)

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in protein synthesis (fractional synthesis rate) in response to eccentric exercise | Up to one week after exercise

CONTACTS AND LOCATIONS:
Locations (1):
- MRC-ARUK Centre of Excellence for Musculoskeletal Ageing Research, Division of Metabolic and Molecular Physiology, Postgraduate Entry Medical School, Royal Derby Hospital, Derby, Derbyshire, United Kingdom